CLINICAL TRIAL: NCT02005081
Title: A Prospective Study Using Actifuse SHAPE Versus Autograft With Demineralized Bone Matrix to Achieve Bone Fusion in Anterior Cervical Corpectomy (ACC)
Brief Title: Baxter: Actifuse SHAPE vs DBX in ACC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Hazem Eltahawy MD, Assistant Professor, Neurosurgeon, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Baxter
Record Dates: First submitted 2013-11-01; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Cervical Spine Degenerative Disease Nos; Cervical Spondylosis With Myelopathy
MeSH Terms: interventions — Transplantation, Autologous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Actifuse SHAPE (Other): Actifuse Synthetic Bone Graft substitutes mixed with bone marrow aspirate in cervical spine fusion. Actifuse is a synthetic, porous, silicate-substituted hydroxyapatite and has shown that this maximizes a favorable bony response.
  Interventions: Device: Actifuse SHAPE
- Autograft with Demineralized Bone Matrix (Other): autograft mixed with demineralized bone matrix in cervical spine fusion.
  Interventions: Device: Autograft with Demineralized Bone Matrix

INTERVENTIONS:
Device: Actifuse SHAPE — Actifuse Synthetic Bone Graft substitutes mixed with bone marrow aspirate in cervical spine fusion. Actifuse is a synthetic, porous, silicate-substituted hydroxyapatite and has shown that this maximizes a favorable bony response.
  Arms: Actifuse SHAPE
Device: Autograft with Demineralized Bone Matrix — autograft mixed with demineralized bone matrix in cervical spine fusion.
  Arms: Autograft with Demineralized Bone Matrix

SUMMARY:
The purpose of this single-center, prospective, randomized study is to determine the fusion rates along with the clinical outcomes of commercially available bone graft substitutes Actifuse mixed with bone marrow aspirate (BMA) versus autograft mixed with demineralized bone matrix (DBM), in subjects who require anterior cervical corpectomy (ACC) spinal fusion in patients experiencing cervical spondylotic myelopathy (CSM).

DETAILED DESCRIPTION:
Background Fusion of the spine was introduced in 1911 for the management of deformity and is currently used to relieve pain and restore function in patients diagnosed with degenerative disc disease. Degenerative conditions of the spine resulting in functionally limiting back pain or neck, and arm pain with or without extremity pain and dysfunction are a major problem in today's world. Recommended treatment for these conditions can vary initially from bed rest, exercise, traction, manipulation and drug therapy to eventual surgery.

One of the most common neck conditions that occurs among people older than 50 years is cervical spondylotic myelopathy (CSM). This may produce symptoms of cervical radiculopathy, myelopathy, or both. Over time, the normal wear-and-tear effects of aging can lead to a narrowing of the spinal canal. This compresses or squeezes the spinal cord. CSM can cause a variety of symptoms, including pain, numbness, and weakness. When patients with degenerative cervical disease require surgery, an anterior decompression of the neural elements and reconstruction of the anterior column with allograft, bone graft substitutes or autograft is common. These types of reconstruction surgery can be referred to as Spinal fusion. The objective of spinal fusion is to eliminate motion of the vertebral body and thereby relieve pain.

An anterior cervical corpectomy, fusion and instrumentation, is usually performed for patients who have pressure on their nerves or spinal cord in their neck. This pressure can lead to pain, weakness or numbness in the arms and occasionally in the legs as well. If non-operative treatment such as medications and therapy are ineffective, patients may require surgery in order to relieve the pressure off their spinal cord and nerves.

Anterior cervical corpectomy (ACC) and fusion is performed for patients with symptomatic, progressive cervical spinal stenosis and myelopathy. It is performed to remove the large, arthritic osteophytes (bone spurs) that are compressing the spinal cord and spinal nerves. However, in order to do so generally involves removing nearly the entire vertebral body and disc, which must be replaced with a piece of bone graft or bone graft substitute and mended (fused) together to maintain stability.

Neurosurgeons and orthopedic surgeons are performing bone grafting procedures more frequently. Surgical applications include treating bone defects, fracture fixation, spinal fusion and in the revision of failed total joint arthroplasties. According to data collected by the American Academy of Orthopedic Surgeons, more than 500,000 bone graft procedures are performed annually in the United States.

The most common source of bone graft used to be autograft, the transfer of a small piece of the patient's own bone from one site, usually the iliac crest, to another. However, the amount that can be harvested safely is limited; it increases surgery time and may be complicated by donor site morbidity. The use of allograft, supplying bone graft from other patients via bone banks, overcomes these difficulties. However, the demand for allograft now exceeds the supply, there is a small but finite risk of disease transmission, and it is highly variable in strength. These factors have led to increasing interest in the use of synthetic bone graft substitutes.

This study will assess the fusion rates along with the clinical outcomes for the use of Actifuse Synthetic Bone Graft substitutes mixed with bone marrow aspirate and autograft mixed with demineralized bone matrix in cervical spine fusion. Actifuse is a synthetic, porous, silicate-substituted hydroxyapatite and has shown that this maximizes a favorable bony response.

Study Design This randomized study will be conducted prospectively. The clinical and radiological outcomes of subjects undergoing anterior cervical corpectomy will be documented. There will be a total of 40 subjects enrolled, 20 in each arm - Actifuse with BMA versus autograft with DBM. It is anticipated that the study length will be 42 months this is based on a recruitment period of 18 months followed by a 24 month post-operative follow-up period for each patient included in the study. Subjects will be randomized 1:1 per arm. Randomization will be established at the study site by sealed envelopes accessed at the time of surgery. The sample size of 40 patients will allow statistical comparison between the 2 arms based on a postulated fusion rate of 85 %. Given that this is a single center study with recruitment over 18 months, the total of 40 subjects is a reasonable goal.

Patient Population Subjects enrolled in this study will be identified from the surgeon's medical practice and will include subjects who have failed conservative treatment and have been identified by their own physician as requiring anterior cervical corpectomy, fusion and instrumentation.

Subjects will be suffering from symptoms with the primary diagnosis of cervical spondylotic myelopathy or cervical spinal stenosis in one to four contiguous levels between C3 and T1.

Data Collection The clinical site's research coordinator or nurse will complete case report forms. Data will be collected prospectively, after the patient has agreed to participate in the study by signing the consent form. Data will be collected from the patient's medical records, departmental based electronic records and radiographic reports to verify eligibility. Once the patient is verified eligible for the study, data will be collected from the same sources above. Information will be captured on case report forms. The patient will also complete questionnaire forms. The information collected will be used for study analysis results.

Parameters To Be Assessed Demographics, medical history, X-ray results, quality of life (SF-36), CT Scan results, Concomitant medications, adverse events, pregnancy test, Body Mass Index (BMI), Concomitant therapies, diagnosis, comorbidities, fusion rate, visual analogue scale (VAS) for pain, Neck Disability Index (NDI) Questionnaire, Neurological examination results, clinical assessments and device malfunction, type and duration of surgery, OR room time, bone graft details, blood loss, length of hospital stay (LOS),return to work, revision surgeries and complications.

ELIGIBILITY:
Inclusion Criteria:

* The subject has failed conservative treatment and is a candidate for spinal fusion surgery.
* The subject is ≥18 years old and of legal age of consent.
* The subject is, in the investigator's opinion, psychosocially, mentally, and physically able to fully comply with this protocol, including the post-operative regimen, attend the required follow-up visits, completion of required forms, and be able to understand and provide written informed consent.
* The subject is skeletally mature (epiphyses closed).
* The subject has voluntarily signed the approved informed consent.
* The subject is willing and able to participate in post-operative clinical and radiographic follow up evaluations for 2 years.
* No previous surgical intervention at the involved fusion level(s);
* Women of child-bearing potential must not be pregnant or nursing, and agrees to not get pregnant for 1 year following surgery

Exclusion Criteria:

* Subject has systemic infection or infection at the surgical site.
* Subject has a medical condition that would interfere with post-operative assessments and care (i.e., metabolic bone disease, neuromuscular disease, autoimmune disease, active malignancy, psychiatric disease, paraplegia, quadriplegia, etc.).
* Subject has a concurrent disease process that would place the subject in excessive risk to surgery (i.e. significant circulatory or pulmonary problems, or significant cardiac disease).
* Subject has a history (present or past) of substance abuse (recreational drugs, prescription drugs or alcohol) that in the investigator's opinion may interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow-up.
* The subject is pregnant/breastfeeding at the time of enrollment, or plans to become pregnant during the course of the study.
* Subject is participating in another clinical study, which could confound results.
* Subject has ossification of posterior longitudinal ligament (OPLL) at any level
* History of an osteoporotic fracture of the spine, hip or wrist
* History of an endocrine or metabolic disorder (e.g., Paget's disease) known to affect bone and mineral metabolism
* Taking medications that may interfere with bony/soft tissue healing including chronic steroid use
* Known allergy to titanium, stainless steels, polyurethane, polyethylene, or ethylene oxide residuals
* Rheumatoid arthritis or other known autoimmune disease or known to have a systemic disorder such as HIV, active hepatitis B or C or fibromyalgia
* Severe obesity (Body Mass Index > 40)
* Physical or mental condition (e.g., psychiatric disorder, senile dementia, Alzheimer's disease, alcohol or drug addiction) that would interfere with patient self-assessment of function, pain or quality of life.
* Involved in current or pending spinal litigation where permanent disability benefits are being sought
* Incarcerated at the time of study enrollment
* Diseases that significantly inhibit bone healing (osteoporosis, metabolic bone disease, uncontrolled diabetes, dialysis dependent renal failure, symptomatic liver disease)
* Undergoing chemotherapy or radiation treatment, or chronic use of steroids (defined as more than 6 weeks of steroid use within 12 months of surgery, other than episodic use or inhaled corticosteroids)
* Subject has severe osteopenia, osteoporosis, osteomalacia, spinal metastases, or metabolic bone disease that would significantly inhibit bone healing OR the level of BMD is a T score of -2.5 or below OR patient has sustained a vertebral compression or nontraumatic hip or wrist fracture.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Change in Fusion Rates | Baseline, 6 weeks, 6 months, 12 months, 24 months
  2 or 4 view x-rays (Lateral, Flexion, Extension, Anteroposterior)at 6 weeks, 6 months, 12 months and 24 months CT scan at 12 months and 24 months Radiographic Fusion Success is defined as evidence of:Bridging trabecular bone on two contiguous segments in two or three planes (axial, sagittal, or coronal),Translational motion less than 3 mm as measured on flexion/extension films,Angular motion less than 3 degrees as measured on flexion/extension films Note: For multi level fusions, all levels must be fused according to the above criteria.
  Reported at study completion.

SECONDARY OUTCOMES:
Change in Clinical Outcomes | Baseline, 6 weeks, 6 months, 12 months and 24 months
  Pain/Function Disability Subjects must exhibit an improvement compared to their preoperative scores in the following measures to be considered a success:Neck Disability Index (NDI),Visual Analogue Scale (VAS),Quality of Life (SF-36v2 - 1 week recall)
  Reported at study completion.
Change in Clinical Outcomes | Baseline, 6 weeks, 6 months, 12 months, 24 months
  Neurological Status Subjects will be considered to be a neurological success if they experience maintenance or improvement of their neurological status when compared to baseline scores.
  Reported at study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Hazem Eltahawy, MD, Principal Investigator — Wayne State University, DMC
Locations (1):
- Wayne State University, Detroit, Michigan, United States